CLINICAL TRIAL: NCT01945554
Title: The Value of Short-term Pain Relief for the Prediction of Long-term Outcome After Cervical or Lumbar Nerve Root Infiltration
Acronym: InfStu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holger Joswig (Other)
Responsible Party: Sponsor-Investigator, Holger Joswig, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 13/061
Record Dates: First submitted 2013-09-10; First posted 2013-09-18 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cervical Disc Herniation; Lumbar Disc Herniation
Keywords: infiltrative therapy; cervical disc herniation; lumbar disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Bupivacaine; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical disc herniation (Experimental): Patients with cervical disc herniation and compression of nerve roots C3-C8.
  Interventions: Procedure: Cervical nerve root infiltration; Drug: Mephamesone; Drug: 0.5% bupivacaine (Bupivacain®)
- Lumbar disc herniation (Experimental): Patients with lumbar disc herniation and compression of nerve roots L1-S1.
  Interventions: Procedure: Lumbar nerve root infiltration; Drug: 0.5% bupivacaine (Bupivacain®); Drug: Kenacort®

INTERVENTIONS:
Procedure: Cervical nerve root infiltration — 4mg Mephamesone followed by 1ml of 0.5% bupivacaine (Bupivacain®) will be administered.
  Arms: Cervical disc herniation
Procedure: Lumbar nerve root infiltration — 40mg triamzinolone (Kenacort®) followed by 2ml of 0.5% bupivacaine (Bupivacain®) will be administered.
  Arms: Lumbar disc herniation
Drug: Mephamesone
  Arms: Cervical disc herniation
Drug: 0.5% bupivacaine (Bupivacain®)
Drug: Kenacort®
  Arms: Lumbar disc herniation

SUMMARY:
The purpose if this study is to assess the response to nerve root infiltration therapy in patients with cervical or lumbar disc herniations.

DETAILED DESCRIPTION:
This prospective, observational study examines the response to routine infiltration therapy in patients suffering from disc herniations of the spine. Using health-related quality of life questionnaires (SF-12 and Neck Pain and Disability Scale and Oswestry Disability Index) and the visual analogue scale the patients will be categorized into ultra-early-, early-, mid-term-, late-responders and non-responders. A two year follow-up of up to 250 patients is planned. With the anonymized participation of this study no patient will experience a change in his treatment plan. Valuable therapeutic management considerations might be drawn from the published results of this study for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic (pain) one-level cervical (C3-C8) or lumbar (L1-S1) radiculopathy with radiological evidence of discal nerve root compression
* Minimum VAS of 20/100
* Age between 18 - 70 years

Exclusion Criteria:

* Multilevel disc herniations with multiple symptomatic nerve root compressions
* Higher motor deficits (Paresis M 0-3 of a peripheral muscle)
* Age < 18 or > 70 years
* Pregnancy
* Allergic reaction against steroids or local anaesthetic
* Bleeding disorder (Tc < 100.000/ul, Quick <50%, INR > 1.5, abnormal PTT)
* Known bleeding diathesis
* Continued anticoagulants (Warfarin = Marcoumar must be bridged with low- or high-molecular heparin; commonly, intake of Aspirin or Clopidogrel is no contraindication for infiltration therapy but is routinely paused when possible)
* Pseudoradicular pain (e.g. in facet arthrosis, iliosacral arthrosis...) - as evaluated to the best of the knowledge of the admitting physician and radiologist performing the infiltration
* Osseous spinal or foraminal stenosis
* Myelopathy
* Severe scoliosis
* Active neoplasm
* History of spinal infection / spondylodiscitis
* History of spinal surgery or previous infiltration therapy on the currently painful segment
* Rheumatic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | 1 month
  (SF)-12 questionaire Change from Baseline SF-12 at 1 month

SECONDARY OUTCOMES:
Neck Pain and Disability Scale (NPAD) | Before, 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Neck Pain and Disability Scale (NPAD)
Oswestry Disability Index (ODI) | Before, 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Oswestry Disability Index (ODI)
Percent change of pain (VAS) | Before, 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Percent change of pain (VAS)
Need for additional surgical therapy and time-to-surgery. | 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Need for additional surgical therapy and time-to-surgery.
Need for hospitalization for disabling pain and time-to-hospitalization. | 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Need for hospitalization for disabling pain and time-to-hospitalization.
Need for repeated infiltrations and time-to-infiltration between the study groups. | 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Need for repeated infiltrations and time-to-infiltration between the study groups.
Absolute VAS pain reduction of a repeated "boost"-infiltration | 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Absolute VAS pain reduction of a repeated "boost"-infiltration
Frequency of opioid use (yes/no) | Before, 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Frequency of opioid use (yes/no)
Ability to return to work (0-100%) and time-to-return to work. | Before, 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Ability to return to work (0-100%) and time-to-return to work.
Health-related quality of life (HRQoL) | Before, 14 days, 1, month, 3 months, 6 months, 12 months, 24 months
  (SF)-12 questionaire
Reasons for 2nd infiltration / surgery | 1 month, 3 months, 6 months, 12 months, 24 months
  Reasons may be either pain and/or sensory dysfunction and/or motor weakness
Patient's satisfaction with therapy | 14 days, 1 month, 3 months, 6 months, 12 months, 24 months
  Would you opt for an infiltration again (provided you had the same outcome as now)?
  * certainly yes
  * maybe yes
  * unsure
  * maybe no
  * certainly no

CONTACTS AND LOCATIONS:
Overall Officials: Holger Joswig, M.D., Principal Investigator — Cantonal Hospital St. Gallen, Dept. of Neurosurgery
Locations (3):
- Switzerland (3):
  - Flawil Hospital, Flawil, Canton of St. Gallen
  - Rorschach Hospital, Rorschach, Canton of St. Gallen
  - Cantonal Hospital St. Gallen, Sankt Gallen